CLINICAL TRIAL: NCT04607902
Title: Harnessing Network Science to Personalize Scalable Interventions for Adolescent Depression: Do Idiographic Symptom Structures Predict Response to Single Session Interventions?
Brief Title: Harnessing Network Science to Personalize Scalable Interventions for Adolescent Depression (TRACK to TREAT Phase 2)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Jessica Schleider, Assistant Professor of Psychology, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB2019-00382
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Depression
Keywords: Single Session Intervention; Online Intervention; Adolescent Depression; Mood Disorders; Experience Sampling Method
MeSH Terms: conditions — Depression; Mood Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (via a random number generator in Qualtrics, double-masking the randomization procedure) to one of the conditions.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized to the Behavioral Activation SSI (BA-SSI), Growth Mindset SSI (GM-SSI), or the Supportive Therapy SSI (ST-SSI; each 30 minutes in length).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supportive Therapy SSI (ST-SSI) (Active Comparator): The web-based supportive therapy (ST-SSI) intervention, called the Sharing Feelings Intervention, is designed to mimic supportive therapy (ST). The goals of the ST intervention are to encourage participants to identify and express feelings to close others; the intervention does not teach or emphasize specific skills or beliefs. In previous clinical trials, ST has resulted in significantly fewer reductions in youth internalizing problems compared to cognitive-behavioral and growth mindset interventions. The ST-SSI is designed to control for nonspecific aspects of intervention, including engagement in a computer program. It includes the same number of reading and writing activities as the other SSIs.
  Interventions: Behavioral: Supportive Therapy SSI
- Behavioral Activation SSI (BA-SSI) (Experimental): The BA-SSI include 5 elements: (1) An introduction to the program's rationale: that engaging in value-based activities can combat sad mood and low self-esteem; (2) Psychoeducation about depression, including how behavior shapes feelings and thoughts; (3) A life values assessment, where youth identify key areas from which they draw enjoyment and meaning; (4) Creation of an activity hierarchy, where youth identify and personalize (in guided exercises) 3 activities to target for change; and (5) An exercise in which youths write about benefits that might result from engaging in each activity; an obstacle that might keep them from doing the activities; and a strategy for overcoming identified obstacles.
  Interventions: Behavioral: Behavioral Activation SSI
- Growth Mindset SSI (GM-SSI) (Experimental): Program includes: An introduction to the brain and a lesson on neuroplasticity; Testimonials from older youths who describe their views that traits are malleable Further stories by older youths, describing times when they used "growth mindsets" to persevere during social/emotional setbacks; Study summaries noting how/why personality can change; And an exercise in which youths write notes to younger students, using scientific information to explain people's capacity for change.
  Interventions: Behavioral: Growth Mindset SSI

INTERVENTIONS:
Behavioral: Supportive Therapy SSI — Online, 30-minute self-administered program for youth
  Other Names: Sharing Feelings SSI; ST-SSI
  Arms: Supportive Therapy SSI (ST-SSI)
Behavioral: Behavioral Activation SSI — Online, 30-minute self-administered program for youth
  Other Names: Activate Action; BA-SSI
  Arms: Behavioral Activation SSI (BA-SSI)
Behavioral: Growth Mindset SSI — Online, 30-minute self-administered program for youth
  Other Names: Project Personality; GM-SSI
  Arms: Growth Mindset SSI (GM-SSI)

SUMMARY:
We will recruit 216 subjects meeting the eligibility criteria. After completing a baseline battery session via secure video conferencing and 3-week phone survey period, adolescents will be randomly assigned to receive 1 of 3 web-based single session interventions (SSIs) at a second secure video conference session. This second session for the intervention will take place within 2-3 weeks after the phone survey period. Immediately pre- and post-SSI, adolescents will complete a limited number of self-report questionnaires to index shifts in proximal outcomes. Participants, both adult and youth, will complete additional follow-up questionnaires 3, 6, 12, 18, and 24 months post-intervention. Participants will complete the intervention, including the pre- and post- SSI questionnaires, and follow-up surveys on their own.

DETAILED DESCRIPTION:
216 eligible adolescents, along with one accompanying parent, will complete a Qualtrics baseline battery via a secure video-conference platform. This battery will be followed by a 3-week (ESM) period. In preparation for this 3-week period, adolescents with a personal smartphone will be assisted in downloading the ecological sampling method (ESM) app during the initial lab session. The participants will then receive an ESM tutorial, and a research team member will review each survey question with the adolescent to ensure comprehension. At the end of the initial session, participating families will schedule a second, brief meeting with the lab to help the adolescent set up the online intervention, which will be completed after the ESM period.

During the ESM period following the baseline battery, adolescents will be prompted to complete the same 2-minute, 8-item survey 5 times per day for 21 days, via a smartphone-based, encrypted data collection app (LifeData). Notifications to complete surveys will occur every 2-3 hours. Responses will be deemed valid if completed within 2 hour of notification, ensuring at least 1-hour lags between surveys.

Once the 3-week ESM period is complete, adolescents will be randomly assigned to receive 1 of 3 web-based single session interventions (SSIs) at a second secure video conference session. The second video conference session will be brief and is meant to help adolescents access the online intervention, which they will complete by themselves. This second session will take place within 2-3 weeks after the ESM period. Immediately pre- and post-SSI, adolescents will complete a limited number of self-report questionnaires by themselves to index shifts in proximal outcomes.

The adolescent and parent pairs will, on their own, complete follow-up assessments at post-intervention. These assessments are abridged versions of the baseline battery. To enable longitudinal analysis of outcome trajectories, adolescents and parents will complete online follow-up questionnaires (including subjective reports of clinical and functional outcomes) 3, 6, 12, 18, and 24 months post-intervention. All follow-up surveys will be completed via Qualtrics, through personalized links sent to the family.

All families will be debriefed by email, and the intervention SSI condition assignment will be revealed, after 24-month follow-up is complete. At this time, adolescents will be offered the opportunity to remotely complete the SSIs they did not originally receive.

ELIGIBILITY:
Inclusion Criteria:

* Ages 11-16 (inclusive) at the time of study enrollment
* Has one parent or legal guardian willing to participate in the study
* Speaks English well enough to complete the smartphone-based questionnaire
* Comfort with smartphone-based surveys
* Indication of elevated risk for youth depression, one of two ways (or both ways): (a) elevations in depressive symptoms, at least 80th percentile or higher, based on parent-report CDI 2; (b) received treatment for depression within the previous 2 years

Exclusion Criteria:

* Fail to meet the above-listed inclusion criteria
* Exit the study prior to condition randomization
* Respond with either copy/pasted responses from text earlier in the intervention to any of free response questions
* Obvious lack of English fluency in open response questions
* Responding with random text in open response questions
* Duplicate responses from the same individual in baseline or follow-up surveys
* Provide responses of fewer than 3 words to writing prompts that ask for at least 2 sentences or more

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in adolescent depressive symptom severity | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  The Children's Depression Inventory (CDI) 2 - short form (CDI-SF) is a reliable, valid measure of youth-reported depression severity, normed for youth age and sex and yielding raw and T scores.

SECONDARY OUTCOMES:
Changes in parent-reported adolescent symptom severity | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  The Children's Depression Inventory (CDI) 2 - parent form will be used to note differences in youth depression severity.

OTHER OUTCOMES:
Demographics | Pre-intervention only (sex, race); Pre-intervention, 3-month follow-up, 6-month follow-up, 12-month follow-up, 18-month follow-up, 24-month follow-up (age, gender identity, mental health treatment history)
  Parents will report demographic, family, and other background information (e.g. age, sex, gender identity, race, mental health treatment history).
Pubertal development | Pre-intervention only
  Youth will complete the Pubertal Development Scale, given effects of puberty on depression onset.
Adverse Childhood Experiences (ACEs) for parent and child | Pre-intervention only
  The ACEs questionnaire will ask parents about their child's and their own exposure to violence, childhood emotional, physical, or sexual abuse, and household dysfunction during childhood.
Self-Hate and related constructs | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  Adolescents' self-hate will be assessed using the 7-item Self-Hate Scale (SHS). Adolescents will indicate the extent to which each statement is true for them (e.g. "I hate myself") on a 7-point Likert scale. The SHS is a valid measure of self-hate, with excellent internal consistency.
Inventory of Depression and Anxiety Symptoms (IDAS-II) | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  Adolescents will complete the 99-item version of the IDAS-II. Respondents indicate the extent to which they had experienced each symptom "during the past two weeks, including today" on a 5-point scale ranging from not at all to extremely. The IDAS contains scales evaluating levels of Dysphoria; Well-Being; Panic; Suicidality, Lassitude, and Insomnia; Social Anxiety and Ill Temper; Traumatic Intrusions scale; and Appetite Loss and Appetite Gain; and Depression and Dysphoria. The IDAS-II is well-validated and nationally-normed for use with adolescents.
Screen for Child Anxiety and Related Disorders (SCARED) | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  Given high comorbidity between depression and anxiety, adolescent anxiety symptom severity will be assessed via adolescent and parent reports using the SCARED: a reliable, valid, widely used youth anxiety assessment with analog parent and youth-report forms.
Behavioral Activation for Depression Scale (BADS)-Short Form | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  Youths' approach versus disengagement from rewarding activities will be assessed via the BADS, a 9-item youth-report questionnaire with strong reliability, predictive validity, and sensitivity to change following BA for adolescent MD.
Self-Referential Encoding Task (SRET) | Pre-intervention
  The SRET is a web-based behavioral measure of self-referent information processing biases that assesses judgements of self-descriptiveness, response latencies and free recall of emotionally valanced stimuli. Adolescents will make decisions about whether positive and negative adjectives are self-descriptive. Participants view various adjectives (26 positive adjectives, 26 negative adjectives) one at a time and make rapid judgments about whether or not each word presented described themselves following word offset. Participants will be told to use the Q or P keys on their keyboard to answer whether the word described them or not. Each trial will be followed by a 1,500 ms intertrial interval.
The Dietary Restriction Screener (DRS) | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  The DRS-2 is a 9-item measure evaluating restrictive eating, bingeing, and purging behaviors in participants. 6 items ask adolescents whether or not they have engaged in restrictive eating, bingeing, or purging behaviors in the past year or in the past 3 months (0 = no; 1 = yes). The other 3 items assess the frequency of these behaviors over the past 28 days.
Self-Injurious Thoughts and Behaviors Interview-Short Form (SITBI-SF) | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  Four items from a self-report version of the SITBI-SF will be used to assess each adolescent's lifetime history of suicide ideation, suicide attempts, and deliberate self-harm. The SITBI-SF is a widely used measure of the continuum of suicidality and self-harm and has demonstrated high test-retest reliability, high internal consistency, and moderate-to-high concurrent validity. Score range for this measure can range widely (per wide variation in instances of self-harming behaviors across one's lifetime); thus, we anticipate a minimum score of 0 and are unable to predict the top (maximum) score.
Secondary Control Scale for Children (SCSC) | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  The SCSC is a 20-item scale measuring youths' perceived ability to shape the personal impact of objective conditions on oneself, by adjusting oneself to fit those conditions. Youth rate agreement with items reflecting various kinds of secondary control, such as adjusting cognition ("When something bad happens, I can find a way to think about it that makes me feel better"). The SCSC has shown acceptable reliability and validity in a large youth sample.
Hopelessness | Immediately Pre- to Immediately Post-intervention; Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  The Becks Hopelessness Scale (BHS) asks both parents and youth to rate 4 statements based on their sense of hopelessness. Participants rate the 4 statements on a 4 point scale ranging from 0 (Absolutely Disagree) to 3 (Absolutely Agree). Total score ranges from 0 to 12, with higher scores indicating greater levels of hopelessness.
Perceived agency | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  The Primary Control Scale for Children (PCSC) is a 24-item scale measuring youths' perceived ability to influence or alter objective events or conditions through personal effort. Youth rate agreement with statements about their ability to exert primary control (e.g., "I can do well on tests if I study hard"; "I can get other kids to like me if I try"). This PCSC has shown acceptable internal consistency, 6-month test-retest reliability, and strong inverse relations to adolescent depressive symptoms.
Implicit Personality Theory Questionnaire (IPTQ) | Immediately Pre- to Immediately Post-intervention; Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  The IPTQ asks youth to rate the extent of their agreement with three statements linked to the malleability of personality, using a 1-to-7 Likert scale (e.g. "Your personality is something about you that you can't change very much." Higher summed scores on these three items indicate a stronger fixed personality mindset, a lower scores, a stronger growth personality mindset.
Brief Family Assessment Measure (General Scale) | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  The BFAMG provides an overview of family functioning. Adolescents and parents rate 14 statements describing the family (e.g. "We feel loved in our family.") using a 0-3 Likert scale.
Multidimensional Peer Victimization Scale | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  The MVPS is a self-report scale assessing adolescents' experiences of peer victimization. This study will include the social manipulation, verbal victimization, and physical victimization scales, totaling 12 items. Adolescents rate how often peers have victimized them in various ways in the past year (e.g. "called me names"; "tried to turn my friends against me").
UCLA Loneliness Scale | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  The ULS is a widely used self-report scale of loneliness in adolescents. The brief 8-item version will be used here. Adolescents rate agreement with 8 items reflecting loneliness (e.g. "I feel left out"; "I feel isolated from others"). The ULS has shown adequate reliability and validity in adolescent samples.
Brief Symptom Inventory-18 | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  The BSI-18 is a valid, reliable screening tool for adult (here, parental) psychological distress. Adult respondents rate endorsement of 18 physical and emotional complaints on a 0-4 Likert scale. The BSI-18 includes 3 subscales for somatic, anxiety, and depressive symptoms, respectively. The total sum score yields an additional total distress score.
Perceived barriers to treatment | Pre-SSI only
  Parents will complete the Barriers to Accessing Care Evaluation at baseline, modified for use by parents. Parents rate the degree to which various beliefs, concerns, circumstances, and logistical difficulties have stopped, delayed or discouraged them from getting professional care for their child's mental health problem. Higher total scores indicate greater perceived barriers to care.
Prognostic Pessimism For Depression | Pre-intervention to 3-month follow-up; Pre-intervention to 6-month follow-up; Pre-intervention to 12-month follow-up; Pre-intervention to 18-month follow-up; Pre-intervention to 24-month follow-up
  Prognostic Pessimism for Depression (PPD) consists of five short questions, adapted from previous research, that aim to quantify a participants' perception of depression as a fixed or malleable condition. Both parents and adolescents will complete the PPD. Questions ask how permanent participants expect depression to be, why, and what might make it less so. An analogous set of questions are posed to parents, who are asked to respond about their children.
COVID-19 Items | Pre-intervention only
  Adapted from CDC Item Bank questions, these questions ask parents about the effects of COVID-19 on their families. Questions ask about stress caused by the pandemic, coping, illness, and effects on other items such as finances, mental health treatment, and employment.
Ecological Sampling Method Surveys (ESM) | Pre-intervention only
  The ESM surveys will include selected items from the Patient Health Questionnaire-9, a widely-used measure of adolescent and adult depressive symptoms. Items will assess symptoms that could plausibly shift in any 2-3 hour period. At the end of the final survey on each day, adolescents will be asked two additional free response questions: "What was the most pleasant event today?" and "What was the most unpleasant event today?".

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Schleider, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The data and protocol from this study will be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After study completion
Access Criteria: Open to public